CLINICAL TRIAL: NCT06304805
Title: A Randomized, Open-label, Single-dose, 3-cycle, 6-sequence, Crossover Study Evaluating Food Effect on Pharmacokinetic Profiles of TGRX-326 in Chinese Healthy Subjects and Effect of Drug Specification on Bioavailability in Human
Brief Title: TGRX-326 Pharmacokinetic Food Effect Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TGRX-326-1002
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a PK assessment study, hence only bio-sample analysis personnel were masked for the type of treatment received for each sample to avoid bias in analysis. Other study personnel, including participants, investigators and staffs were not masked for treatment types.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group A (Experimental): cycle 1: treatment drug + fasted cycle 2: reference drug + fasted cycle 3: treatment drug + food
  Interventions: Drug: cycle 1: treatment drug; Behavioral: cycle 1: fasted; Drug: cycle 2: reference drug; Behavioral: cycle 2: fasted; Drug: cycle 3: treatment drug; Behavioral: cycle 3: food
- Group B (Experimental): cycle 1: reference drug + fasted cycle 2: treatment drug + food cycle 3: treatment drug + fasted
  Interventions: Drug: cycle 1: reference drug; Behavioral: cycle 1: fasted; Drug: cycle 2: treatment drug; Behavioral: cycle 2: food; Drug: cycle 3: treatment drug; Behavioral: cycle 3: fasted
- Group C (Experimental): cycle 1: treatment drug + food cycle 2: treatment drug + fasted cycle 3: reference drug + fasted
  Interventions: Drug: cycle 1: treatment drug; Behavioral: cycle 1: food; Drug: cycle 2: treatment drug; Behavioral: cycle 2: fasted; Drug: cycle 3: reference drug; Behavioral: cycle 3: fasted
- Group D (Experimental): cycle 1: treatment drug + food cycle 2: reference drug + fasted cycle 3: treatment drug + fasted
  Interventions: Drug: cycle 1: treatment drug; Behavioral: cycle 1: food; Drug: cycle 2: reference drug; Behavioral: cycle 2: fasted; Drug: cycle 3: treatment drug; Behavioral: cycle 3: fasted
- Group E (Experimental): cycle 1: reference drug + fasted cycle 2: treatment drug + fasted cycle 3: treatment drug + food
  Interventions: Drug: cycle 1: reference drug; Behavioral: cycle 1: fasted; Drug: cycle 2: treatment drug; Behavioral: cycle 2: fasted; Drug: cycle 3: treatment drug; Behavioral: cycle 3: food
- Group F (Experimental): cycle 1: treatment drug + fasted cycle 2: treatment drug + food cycle 3: reference drug + fasted
  Interventions: Drug: cycle 1: treatment drug; Behavioral: cycle 1: fasted; Drug: cycle 2: treatment drug; Behavioral: cycle 2: food; Drug: cycle 3: reference drug; Behavioral: cycle 3: fasted

INTERVENTIONS:
Drug: cycle 1: treatment drug — for cycle 1 treatment: participants are given the oral treatment specification (60 mg *1 pill)
  Arms: Group A; Group C; Group D; Group F
Drug: cycle 1: reference drug — for cycle 1 treatment: participants are given the oral reference specification (5 mg *2 pills + 25 mg * 2 pills)
  Arms: Group B; Group E
Behavioral: cycle 1: fasted — for cycle 1 treatment: participants are asked to take the drug fasted
  Arms: Group A; Group B; Group E; Group F
Behavioral: cycle 1: food — for cycle 1 treatment: participants are asked to take the drug after food intake
  Arms: Group C; Group D
Drug: cycle 2: treatment drug — for cycle 2 treatment: participants are given the oral treatment specification (60 mg *1 pill)
  Arms: Group B; Group C; Group E; Group F
Drug: cycle 2: reference drug — for cycle 2 treatment: participants are given the oral reference specification (5 mg *2 pills + 25 mg * 2 pills)
  Arms: Group A; Group D
Behavioral: cycle 2: fasted — for cycle 2 treatment: participants are asked to take the drug fasted
  Arms: Group A; Group C; Group D; Group E
Behavioral: cycle 2: food — for cycle 2 treatment: participants are asked to take the drug after food intake
  Arms: Group B; Group F
Drug: cycle 3: treatment drug — for cycle 3 treatment: participants are given the oral treatment specification (60 mg *1 pill)
  Arms: Group A; Group B; Group D; Group E
Drug: cycle 3: reference drug — for cycle 3 treatment: participants are given the oral reference specification (5 mg *2 pills + 25 mg * 2 pills)
  Arms: Group C; Group F
Behavioral: cycle 3: fasted — for cycle 3 treatment: participants are asked to take the drug fasted
  Arms: Group B; Group C; Group D; Group F
Behavioral: cycle 3: food — for cycle 3 treatment: participants are asked to take the drug after food intake
  Arms: Group A; Group E

SUMMARY:
A study evaluating the effects of food intake on the pharmacokinetic (PK) profiles of TGRX-326 and the effect of different drug specifications on human bioavailability for TGRX-326, a drug indicated for non-small cell lung cancer treatment

DETAILED DESCRIPTION:
This study is designed as single-center, randomized, open-label, 3-cycle, 6-sequence and crossover design to evaluate 1) food effect on PK profile of TGRX-326; 2) effect of different specifications of TGRX-326 on human bioavailability. Safety for food effect on TGRX-326 and safety for different TGRX-326 specifications were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* able to understand the purpose, methods and possible adverse events of the study and agree to volunteering consent before the start of study
* healthy subject; male or female
* Age between 18 and 55 (inclusive)
* body mass index (BMI) between 19.0 and 26.0 (inclusive), male weight <=50 kg, female weight <=45 kg
* normal/ clinically insignificant test results (including physical exam, laboratory tests, 12-lead ECG, chest x-ray, etc.)
* participant/partner of the participant does not have plans for child bearing from screening until 6 months after study, and is willing to take contraceptive measures during study period and for 6 months, and does not have plans to donate sperm/egg during the said period

Exclusion Criteria:

* history of allergic reactions, or allergic to any components to the study drugs that by investigator's judgement unsuitable for the study
* any clinically significant conditions that could affect study outcomes, safety or compliance
* history of major surgery within 3 months before first dose, or have plans to receive surgery during the study, or history of any surgery that could affect drug absorption, distribution, metabolism and excretion
* have difficulties to receive venous needle puncture, or cannot tolerate venous needle puncture, or history of hematophobia or needle sickness
* history of substance abuse
* have special food requirement or cannot follow food requirement of the study, or lactose intolerant
* use of any investigational drug or participation of any clinical study (for drug or medical device) within 3 months before first dose, or cannot participate the study in person/on site
* history of blood donation, blood loss (>= 400 mL, excluding normal blood loss during female menstrual period), or reception of blood transfusion within 3 months before screening
* history of daily cigarette consumption of more than 5 within 3 months before screening, or cannot avoid using cigarette/tabacco products during the study
* history of alcohol abuse (more than 14 units of alcohol per week) within 3 months before screening, or cannot avoid alcohol consumption during study
* history of large tea/coffee/caffeinated drink intake (more than 8 cups per day) within 3 months before first dose
* history of irregular dietary schedule within 1 months of first dose (including, dieting, overeating, low sodium intake, etc.)
* use of any prescription / over-the-counter drug, or Chinese herbal medication, or health supplementary products within 14 days of test article administration
* vaccination within 14 days before first test article administration, or have plans to receive vaccination during the study period
* any one positive result for hepatitis-B surface antigen, Hepatitis C antibody, HIV antibody or syphilis antibody
* alcohol breathing test results of > 0.0 mg/100mL for blood alcohol concentration
* positive test results on substance use (including, morphine, methylamphetamine, ketamine, tetrahydrocannabinol, methylene-dioxy-methyl-amphetamine)
* female in pregnancy or breastfeeding period, or positive pregnancy test result
* history of unprotected sexual activities within 14 days before first dose
* consumption of food or drink rich in caffeine/xanthine (such as chocolate, coffee, tea, coke) or food/food product of grapefruit, dragon fruit, mango, tangerine, or any food that could affect drug absorption, distribution, metabolism and excretion
* any reasons that is deemed unsuitable for study participation as determined by investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Plasma Cmax | During treatment period on Day 1 of each of three cycles (each cycle is one day, and there is a 10-day washout period between two cycles)
  Maximum concentration of TGRX-326 measured in plasma
Plasma AUC(0-t) | During treatment period on Day 1 of each of three cycles (each cycle is one day, and there is a 10-day washout period between two cycles)
  Area Under drug concentration-time curve (AUC) from time 0 to last measureable timepoint for TGRX-326 as measured in plasma
Plasma AUC(0-inf) | During treatment period on Day 1 of each of three cycles (each cycle is one day, and there is a 10-day washout period between two cycles)
  Area Under drug concentration-time curve from time 0 to infinity for TGRX-326 as measured in plasma

SECONDARY OUTCOMES:
Plasma Tmax | During treatment period on Day 1 of each of three cycles (each cycle is one day, and there is a 10-day washout period between two cycles)
  Time to maximum concentration of TGRX-326 measured in plasma
terminal elimination rate constant (lambda-z) | During treatment period on Day 1 of each of three cycles (each cycle is one day, and there is a 10-day washout period between two cycles)
  terminal elimination rate constant calculated from plasma TGRX-326 concentrations
Elimination half-life (T1/2-Z) | During treatment period on Day 1 of each of three cycles (each cycle is one day, and there is a 10-day washout period between two cycles)
  Time for TGRX-326 to decrease from maximum plasma concentration to half of maximum plasma concentration
AUC(%Extrap) | During treatment period on Day 1 of each of three cycles (each cycle is one day, and there is a 10-day washout period between two cycles)
  Calculated percentage of Area under curve for AUC(0-inf) that is from last measurable timepoint ot infinity, calculated based on TGRX-326 plasma concentration over time curve.
Plasma volume of distribution (Vz/F) | During treatment period on Day 1 of each of three cycles (each cycle is one day, and there is a 10-day washout period between two cycles)
  Apparent volume of distribution of TGRX-326 in plasma
Plasma clearance (CL/F) | During treatment period on Day 1 of each of three cycles (each cycle is one day, and there is a 10-day washout period between two cycles)
  Apparent clearance of TGRX-326 in plasma
Adverse events/serious adverse events | through completion of the study, a total duration of 37 days
  to record and analyse subjects with adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, MD, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- First Affiliated Hospital Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No